CLINICAL TRIAL: NCT02133053
Title: Non Interventional Study of Ectoin Allergy Nasal Spray Compared to Beclomethasone Nasal Spray
Brief Title: Application of Ectoin Allergy Nasal Spray in Comparison to Beclomethasone Nasal Spray
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PPL-042
Record Dates: First submitted 2014-05-02; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Ectoine; bitop; Ectoin
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Equipment and Supplies; Beclomethasone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ectoin Group: Ectoin Allergy Nasal Spray (Medical Device, drug-like)
  Interventions: Other: Medical Device, drug-like
- Beclomethasone Group: Beclomethasone nasal spray
  Interventions: Drug: Beclomethasone

INTERVENTIONS:
Other: Medical Device, drug-like — Ectoin Allergy Nasal Spray
  Groups: Ectoin Group
Drug: Beclomethasone — Beclomethasone nasal spray
  Groups: Beclomethasone Group

SUMMARY:
This is a comparative, open label, parallel group, non interventional study to further demonstrate the effectiveness and tolerability of Ectoin® Allergy Nasal Spray. In addition the effectiveness and safety shall be compared to a Beclomethasone nasal spray. The patient applies Ectoin® Rhinitis Nasal Spray or Beclomethasone nasal spray according to the instructions for use. The observation takes place over a period of 14 days. Response to treatment is recorded at day 7 and day 14 by the physician and in daily by the patient in a dairy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed allergic rhinitis during the observational period

Exclusion Criteria:

* Contra indications according to the label

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score | Time Frame: day 1, day 7, day 14

SECONDARY OUTCOMES:
Change in palatal itching score | Day 1, 7 and 14
Efficacy and tolerability assessment by the patients and by the investigator | day 7 and 14
Change in quality of life assessed by Rhinitis Quality of Life Questionnaire | Day1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Sonnemann, MD, Principal Investigator — HNO Praxis Elmshorn